

## VALUES AND VIRTUES OF GRANDPARENTS CARING FOR THEIR GRANDCHILDREN AS PROTECTIVE FACTORS OF THEIR HEALTH AND PSYCHOLOGICAL WELLBEING



## STATISTICAL ANALYSIS PLAN

To analyze differences in psychological well-being and quality of life based on sociodemographic variables, **Student's t-tests** and **one-way ANOVA** will be performed. To analyze the relationships between character virtues-strengths, psychological well-being, emotional competencees, quality of life, role satisfaction, and overload and involvement, **Pearson correlations** will be carried out and, subsequently, **regressions** will be performed to find out which virtues (and, more specifically, strengths) and competences have the greatest weight in psychological well-being and quality of life. Finally, **repeated measures ANOVAs** and **ANCOVAS** will be performed to analyze the effectiveness of the program.

For the analysis of the differential efficacy of the programs, Repeated measures analysis of covariance will be performed. As an intersubject factor, the intervention conditions (GT and GC) will be considered and as an intrasubject factor the evaluation phases (pre-intervention, post-intervention and follow-up). The effect of the intervention will be analyzed considering as dependent variable both psychological well-being and quality of life and those which, according to theoretical approaches, are the mechanisms of action through which the intervention is hypothesized to act (e.g. emotional competences, strengths). Depending on the results obtained in other variables and on the possible difference between pre-intervention conditions in some of these variables, the inclusion of covariates will be considered. In particular, statistically significant results are expected to be obtained when analyzing the interaction between the change associated with the interventions and the passage of time, since this measure will indicate the extent to which the scores between the two groups (intervention and control) differ in the post-intervention and follow-up phases. Differences will be analyzed according to the gender of the participants.

In addition, an Intention-to-treat analysis will be performed so that all grandparents who initiate treatment will be included in the analyses of the efficacy of the intervention. That is, all subjects who initiate treatment will be included in the analyses. Thus, in the case of dropouts, all data from their last recorded time of measurement will be maintained in the post-treatment and follow-ups. Values will be kept for pre-treatment when caregivers drop out without completing



treatment and for the last follow-up when they drop out once treatment is completed (Kazdin, 1998).

Following the recommendations of the American Psychological Association (APA), the effect size of the results obtained will be analyzed. In addition to the analysis of the results in terms of whether statistically significant changes associated with the intervention occur, an analysis of the clinical significance of such changes will be conducted. The assessment of whether significant clinical changes occur over time for each grandparent will be performed through the procedure outlined by Jacobson et al. (1999), through which a score (reliable change index) is obtained which, if greater than 1.96, indicates that a clinically significant positive change in the score has occurred, while if less than -1.96 indicates that a clinically significant negative change in the score has occurred. Scores between 1.96 and -1.96 indicate that no significant change has occurred as a result of the intervention.

The evaluation of the program will be carried out following the program assessment methodology. The program content, the implementation process, the results obtained and the impact generated will be evaluated. The resources to be used will include documents (records, meetings and protocols) and staff (participants, trainers and indirect agents). Data collection techniques will consist of self-reports. To evaluate the program, criteria for implementation, results and outcomes will be established. The process will be considered during the implementation phase. The results will include the achievement of objectives, as well as the satisfaction levels of the participants.